CLINICAL TRIAL: NCT04494373
Title: A Randomized, Double-blinded and Parallel Study to Assess the Pharmacokinetic, Pharmacodynamic, Safety and Immunogenicity of HS-20090 and Xgeva® in Healthy Adults
Brief Title: Comparing of the Pharmacokinetic, Pharmacodynamic, Safety and Immunogenicity of HS-20090 and Xgeva® in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HS-20090-101
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Bone Metastasis From Solid Tumors
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-20090 (Experimental): Subcutaneously injection of HS-20090 (120mg/1.7mL) once on the first day
  Interventions: Drug: HS-20090
- Xgeva® (Active Comparator): Subcutaneously injection of Xgeva® (120mg/1.7mL) once on the first day
  Interventions: Drug: Xgeva®

INTERVENTIONS:
Drug: HS-20090 — A human IgG2 monoclonal antibody with affinity and specificity for human RANKL
  Arms: HS-20090
Drug: Xgeva® — A human IgG2 monoclonal antibody with affinity and specificity for human RANKL
  Arms: Xgeva®

SUMMARY:
A randomized, double-blind and parallel group study to compare the pharmacokinetic, pharmacodynamic, safety and immunogenicity of HS-20090 120mg（1.7ml）and Xgeva® in healthy adults.

DETAILED DESCRIPTION:
This is a phase I, single center, randomized, double-blind and parallel group clinical trial .

The primary objective is to assess the pharmacokinetic similarity of single subcutaneously injection of HS-20090 or Xgeva® in healthy volunteers.

The secondary objectives are to assess the Clinical safety and immunogenicity similarity of single subcutaneously injection of HS-20090 or Xgeva® in healthy volunteers. Meanwhile，observing the pharmacodynamic similarity of HS-20090 to Xgeva® preliminarily.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form and fully understand the test content, process and possible adverse reactions, and be able to complete the study according to the test plan requirements;
* Healthy males, Aged ≥18 years or ≤50 years old(including the boundary value);
* Agree to take effective contraceptive measures throughout the study period until at least 6 months after the last drug is administered;
* Clinical laboratory examination, chest X-ray, abdominal B-ultrasound, electrocardiogram, physical examination, vital signs and various examinations are normal or abnormal without clinical significance.

Exclusion Criteria:

* Occurred or suffering from osteomyelitis or ONJ (mandibular necrosis) previously; The dental or jaw disease that is active, requiring oral surgery; or planned for invasive dental surgery during the study; or dental or oral surgery wounds have not healed;
* Serum calcium levels are outside the normal range of the laboratory.
* Subject has positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result viral hepatitis (including hepatitis B and hepatitis C), or positive HIV antibodies, or positive test for syphilis.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months or 5 half-lives (whichever is longer).
* Prior use of medications within 6 months before and during the study. This includes medications such as, but not limited to: Bisphosphonates Fluoride Calcitonin Strontium Parathyroid hormone or derivatives Supplemental vitamin D (>1000 IU/day) Glucocorticosteroids (topical corticosteroids administered more than 2 weeks prior to enrolment are allowed) Anabolic steroids Calcitriol Diuretics

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC0-t ) | 155days
Cmax | 155days
  maximum concentration

SECONDARY OUTCOMES:
Adverse events(AE) | 155days
  The adverse medical events that occur after the clinical trial subjects receive the test drug do not necessarily have a causal relationship with the treatment.
Serum type 1 C-telopeptide(CTX1) | 155days
  explore the pharmacodynamic profile by detecting the serum concentration of CTX1

OTHER OUTCOMES:
Antidrug antibody(ADA): | 155days
  percentage of subjects positive for antidrug antibody
Neutralizing antibody(Nab) | 155days
  percentage of subjects positive for Nab

REFERENCES:
- [Derived] Lin Y, Yang H, Yang X, Guo C, Yang S, Yang G, Wu Q, Pan C, Sun C, Li C, He L, Huang J, Pei Q. Biosimilarity of HS-20090 to Denosumab in healthy Chinese subjects: a randomized, double-blinded, pharmacokinetics/pharmacodynamics study. Expert Opin Investig Drugs. 2022 Oct;31(10):1125-1132. doi: 10.1080/13543784.2022.2123737. Epub 2022 Sep 16. PMID 36112084